CLINICAL TRIAL: NCT05830305
Title: MOBILE Health Intervention in IntraCerebral Hemorrhage Survivors
Acronym: MOBILE-ICH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Teo Kay-Cheong, Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UW 22-702
Record Dates: First submitted 2023-03-17; First posted 2023-04-26 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Intracerebral Hemorrhage; Hypertension
MeSH Terms: conditions — Cerebral Hemorrhage; Hypertension

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile health intervention (Active Comparator): Subjects will enter their home BP measurements into a mobile stroke App (WeRISE) daily, and the study team will regularly review the BP measurements through a backend system. A protocol-based intervention via phone calls, which includes anti-hypertensive drug adjustment and reinforcement of lifestyle modification, will be implemented.
  Interventions: Other: Mobile health intervention
- Usual care (No Intervention): Subjects will have their hypertension managed by their respective treating physicians.

INTERVENTIONS:
Other: Mobile health intervention — A protocol-based intervention via phone calls, which includes anti-hypertensive drug adjustment and reinforcement of lifestyle modification, will be implemented.
  Arms: Mobile health intervention

SUMMARY:
This randomized controlled trial investigates the efficacy and safety of mobile health intervention in managing hypertension after Intracerebral Hemorrhage (ICH).

DETAILED DESCRIPTION:
140 ICH survivors will be randomized into mobile health intervention (MOBILE) and the usual care group for hypertension management. All subjects will be educated on the importance of hypertension control after ICH and given lifestyle advice, including the DASH diet. Subjects in the MOBILE group will enter their home blood pressure (BP) measurements into a mobile stroke App (WeRISE) daily, and the study team will regularly review the BP measurements through a backend system. A protocol-based intervention via phone calls, which includes anti-hypertensive drug adjustment and reinforcement of lifestyle modification, will be implemented. Subjects in the usual care group will have their hypertension managed by their respective treating physicians. All subjects will be followed up for 26 weeks. The primary and secondary endpoints include the rate of controlled hypertension at 12 and 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Primary ICH Diagnosis
* Age ≥ 18 years
* Discharge Modified Rankin Scale of ≤4

Exclusion Criteria:

* Expected life expectancy of <1 year
* Patient or caregiver does not have access to WeRISE App.
* Patient or caregiver does not know how to use WeRISE App .
* Inability to perform home BP monitoring
* Inability to participate in follow-up activity
* Contraindication for intensive and rapid lowering of blood pressure (Known >70% cerebral vascular stenosis; History of fall, dizziness or syncope due to hypotension; Any other medical condition that is deemed contraindicated for low blood pressure
* Bleeding tendency (Platelet count < 75 x 10^9/L; Known coagulation disorder)
* Severe renal impairment (Estimated glomerular filtration rate using CKD-EPI formula <30 ml/min/1.73m2)
* Severe liver impairment (Child-Pugh C cirrhosis)
* Known contraindication or allergy to two or more anti-hypertensive classes

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Rate of controlled hypertension 12 weeks after ICH | 12 weeks
  Office systolic BP <130 mmHg

SECONDARY OUTCOMES:
Change of BP from recruitment to 12 weeks | 12 weeks
  The difference between BP measurement on recruitment and at 12 weeks
Rate of controlled hypertension 26 weeks after ICH | 26 weeks
  Office systolic BP <130 mmHg
Life Simple 7 Score at 12 and 26 weeks | 12 and 26 weeks
  Score ranging from 0-14 points, with the higher scores indicating better lifestyle health

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Background] Biffi A, Teo KC, Castello JP, Abramson JR, Leung IYH, Leung WCY, Wang Y, Kourkoulis C, Myserlis EP, Warren AD, Henry J, Chan KH, Cheung RTF, Ho SL, Anderson CD, Gurol ME, Viswanathan A, Greenberg SM, Lau KK, Rosand J. Impact of Uncontrolled Hypertension at 3 Months After Intracerebral Hemorrhage. J Am Heart Assoc. 2021 Jun;10(11):e020392. doi: 10.1161/JAHA.120.020392. Epub 2021 May 15. PMID 33998241
- [Background] Teo KC, Keins S, Abramson JR, Leung WCY, Leung IYH, Wong YK, Yeung C, Kourkoulis C, Warren AD, Chan KH, Cheung RTF, Ho SL, Gurol ME, Viswanathan A, Greenberg SM, Anderson CD, Lau KK, Rosand J, Biffi A. Blood Pressure Control Targets and Risk of Cardiovascular and Cerebrovascular Events After Intracerebral Hemorrhage. Stroke. 2023 Jan;54(1):78-86. doi: 10.1161/STROKEAHA.122.039709. Epub 2022 Nov 2. PMID 36321455